## NCT02505984

## **Preventing Postpartum Depression with Intranasal Oxytocin**

**Date of document: 12/27/2024** 

## **Data Analysis**

The final sample size includes 38 eligible women randomly assigned to oxytocin administration (n=18) or placebo (n=20). Missing data were allowed such that 18.59% of the data were missing, with 23 different patterns. Jamshidian and Jalal's non-parametric Missing Completely At Random (MCAR) test indicated that the data was Missing At Random (MAR): Hawkins's test,  $\chi^2_{\text{median}(6)} = 14.33$ ,  $p_{\text{median}} = .026$ , and Anderson-Darlin's rank test,  $T_{\text{median}} = 5.88$ ,  $p_{\text{median}} = .005$ . Missing data was handled by Multiple Imputation (Rubin, 2009) with 50 complete sets. The reported basic results are the pooled outcome of the MI procedure. Before the primary analyses, we examined the normal distribution of all the quantitative study measures using a series of Anderson-Darling normality tests. Basic analyses for study group comparison on outcome measures for each time point were performed using Mann-Whitney U tests.